CLINICAL TRIAL: NCT04437069
Title: Improving Patient and Family Health Using Family-Centered Outcomes and Shared Decision-Making
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Angie Fagerlin, Professor & Chair, Department of Population Health Sciences, University of Utah
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB_00103194
Record Dates: First submitted 2020-05-29; First posted 2020-06-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Patient Decision Aids; Congenital Heart Disease; Congenital Heart Defect
Keywords: values clarification exercise; shared decision making; patient education; patient decision aids; congenital heart disease; congenital heart defect
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Parents randomized using simple randomization into two conditions: one group receives the patient decision aid, and one group receives the patient decision aid and the values clarification exercise. There is no stratified randomization. There are 4 survey time points: 1) Baseline, 2) Post-Viewing of the Decision Aid (or Decision Aid and Values Clarification Exercise), 3) Post-Decision, and 4) Three Months Post-Decision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Care (Control) (No Intervention): Participants will receive standard care and will not view either the Decision Aid or the Values Clarification Exercise
- Decision Aid (Experimental): Participants view the Decision Aid only
  Interventions: Other: Decision Aid
- Decision Aid & Values Clarification Exercise (Experimental): Participants view both the Decision Aid and the Values Clarification Exercise
  Interventions: Other: Decision Aid; Other: Values Clarification Exercise

INTERVENTIONS:
Other: Decision Aid — Participants will view a Decision Aid (delivered as an app) that provides them with information regarding congenital heart disease, as described in the literature. The DA is tailored to the specific diagnosis of the fetus/neonate, so that participants are only viewing information about their baby's specific CHD diagnosis (and not other types of CHD). This is shown using videos and diagrams to clearly explain the defect, what their treatment options are (surgical intervention, comfort care, or termination), and personal stories from other parents who have dealt with the same diagnosis before (including both positive and negative outcomes). The DA was developed according to the International Patient Decision Aid Standards (see http://ipdas.ohri.ca/) (IRS# 14-13332).
  Arms: Decision Aid; Decision Aid & Values Clarification Exercise
Other: Values Clarification Exercise — The Values Clarification Exercise is a process that aids patients in clarifying their values and goals to improve alignment of their preferences with their chosen treatment. It was developed according to the International Patient Decision Aid Standards. It includes ten values that were chosen based on feedback from the parent investigators and clinicians. The ten values are: 1) discomfort to the child, 2) time in the hospital, 3) risk that the child will have impairments, 4) need to provide home medical care, 5) chronic medical care/decisions, 6) financial issues, 7) life in adulthood, 8) impact on the family, 9) beliefs about doing everything medically possible, & 10) life expectancy. Each value has a sliding scale where the user can compare 2 treatment options at a time. They are asked which described situation feels better for them and their family.
  Arms: Decision Aid & Values Clarification Exercise

SUMMARY:
This study is a randomized clinical trial where participants (parents of a fetus or neonate diagnosed with a life-threatening congenital heart disease (CHD)) will randomly be assigned to either receiving a web-based decision aid (DA) alone, or receiving the decision aid that includes a values clarification exercise. Because of the novel use of decision aids in CHD in an acute setting, we will also compare participants receiving the DA in a randomized control trial to a prospective observational population of families faced with similar decisions without a DA (control group). We have designated the Brief Symptom Inventory Global Severity Index of Global Distress 3 months post-birth or death/termination as our primary outcome measure.

DETAILED DESCRIPTION:
The diagnosis of a life-threatening pediatric heart condition impacts both the future of a child and the health and quality of life of the family. Parents of a child with this diagnosis are faced with the stress of comprehending extensive information about the diagnosis and treatment options, and are required to make immediate and profound choices about interventions that will have long-lasting repercussions. To provide the best care at this challenging time, it is crucial to find methods to improve parent-provider shared decision making (SDM) and to encourage the inclusion of both patient-centered and family-centered outcomes. One method commonly used to improve SDM are decision aids (DA). DAs are designed to 1) provide accurate and balanced information; 2) clarify patients' values; and 3) improve SDM skills. A Cochrane review showed that DAs contribute to effective SDM by: 1) increasing knowledge of the diagnosis and treatment options, 2) increasing patient and practitioner participation in SDM, 3) reducing uncertainty and decisional conflict, 4) improving concordance between preference and treatment received, and 5) improving patient-provider communication.

Values clarification exercises (VCE) are occasionally included in DAs to help patients clarify their values about the treatment decision. Although these exercises are often used, they are poorly tested. Previous systematic reviews have failed to identify rigorous research studies to answer questions regarding whether VCE improves patient decision making processes. This project aims to determine the impact of the DA with and without the VCE on longitudinal parent mental health, decision quality and perceptions of patient-provider communication. Specifically, we will test the impact of decision aids (DA vs. no DA, and DA with and without the VCE) on mental health outcomes (e.g., anxiety, complicated grief), decision quality (e.g., quality of the decision, parent-provider communication), and provider experience (e.g., satisfaction with interacting with patients who used the tool). In the development of the DA and VCE, we conducted focus groups and interviews in Utah, Illinois, Washington, D.C, and North Carolina with parents whose fetus/neonate had been diagnosed with complex CHD. The main goal of this study is to determine the impact of the DA with and without the VCE on longitudinal parent mental health, decision quality and provider experience.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose fetus/neonate was diagnosed with a life-threatening CHD that meets eligibility criteria below without restriction based on gender, race, age, or socioeconomic status.
* We will request participation from both parents but will not disqualify families if only one parent participates.
* Eligibility Criteria: Parents whose fetus/neonate was diagnosed with a life-threatening CHD that are offered the choice between intervention and comfort care (and in some cases termination). This is limited to the following diagnoses: Truncus Arteriosus, Pulmonary Atresia with Intact Ventricular Septum, Complex Single Ventricle, Complex Single Ventricle with Heterotaxy, Hypoplastic Left Heart Syndrome (HLHS), and Ebstein's Anomaly of the Tricuspid Valve.

Exclusion Criteria:

* Patients with other types of CHD that are not listed above are not eligible.
* Participants must be 18 years of age or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Brief Symptom Inventory (BSI) Global Severity Index of Global Distress | 1 week post baseline & 3 months post-decision
  The BSI is a validated scale of 53 questions that indicate the degree of stress the participant has experienced within the previous seven days. Answers range in a 5 point Likert scale from 0=not at all to 4=extremely. The scale measures stress, so a lower score is better. Scores are obtained for nine primary symptom dimensions and three global indices of distress.
  The primary comparison is the baseline measurement versus 3 months post-decision measurement. We are looking at how those measurements changed.

SECONDARY OUTCOMES:
Decision Quality - Values | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  Six question scale that measures the values that the participant makes while choosing medical treatment. Answers range in a 6-point Likert scale from 1=most important to 6=not as important. There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Decision Quality - Knowledge | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  27 questions assessing the participant's knowledge of treatment options for CHD. Participants not in the intervention arm will also take this survey for comparison. 21 of the questions use a dichotomous response format (either "true / false" or "yes/no"); 5 questions are multiple choice. All questions are answered with full access to the decision aid (if not in standard care arm) since participants are not meant to test recall. "Better" scores will be measured by how many questions that a participant answers correctly.
Perinatal Grief | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  Measured using the Perinatal Grief Scale which measures grief, coping, and despair following the death of a child. This scale was also adapted for a child who did not die. Answers are on a 5-point Likert scale that ranges from 1=strongly agree to 5=strongly disagree. A higher score would indicate less grief, and would therefore be considered "better".
Brief Symptom Inventory (BSI) Global Severity Index of Global Distress | 1 week Post-Decision Aid, 1 month post-decision
  The BSI is a validated scale of 53 questions that indicate the degree of stress the participant has experienced within the previous seven days. Answers range in a 5 point Likert scale from 0=not at all to 4=extremely. The scale measures stress, so a lower score is better. Scores are obtained for nine primary symptom dimensions and three global indices of distress.

OTHER OUTCOMES:
Combined Outcome Measure for Risk Communication and Treatment Decision Making Effectiveness (COMRADE) | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  COMRADE is validated patient-based outcome measure to evaluate the effectiveness of risk communication and treatment decision making in consultations. There are two sub-scales for risk communication and confidence in decision. It allows for paternalistic, shared or informed choice decision making models. There are 10 questions that are answered on a 5 point Likert scale ranging from 1-strongly disagree to 5=strongly agree. Higher scores are better, as they indicate a stronger understanding from the provider.
Preference for Shared Decision Making | 1 week from Baseline, 1 week post-Decision Aid, & 1 month post-decision
  This scale assesses participants' desire to participate in Shared Decision Making. It is an adaptation of the Degner & Sloan's Control Preference Scale. It is a one item question that asks people if they want to make the decision alone, with their clinician, or have their clinician make it. There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Preparation for Decision Making | 1 week Post-Decision Aid
  Preparation for Decision Making Scale is a validated scale which will assess participants' perspectives of the decision aid's usefulness in preparing them to communicate with their clinicians and for Shared Decision Making. These questions are answered on a Likert scale ranging from 1=not at all to 5=a great deal. A higher score indicates that they are better prepared and, thus, a better outcome.
Decision Self-Efficacy Scale | 1 week from Baseline, 1 week post-Decision Aid, & 1 month post-decision
  11 question survey that measures self-efficacy for performing informed decision making (e.g., getting needed information, asking questions, expressing opinions). Answers range in a 5 point Likert scale from 0=not at all confident to 4=extremely confident. Higher scores are better, as they indicate stronger self-efficacy.
Decisional Conflict Scale | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  A 16-question survey that measures 1) perceptions of uncertainty in choosing options, 2) feelings of having adequate knowledge and clear values, and 3) effective decision making. Answers range on a 5 point Likert scale from 0=strongly agree to 4=strongly disagree. Lower scores are better, as they indicate a stronger knowledge about choice availability.
Decisional Regret | 3 months post-decision
  Decision Regret will be assessed by asking participants to reflect on the decision they made about which treatment option they chose for their child. The measure consists of 5 items assessed on a 5-point Likert scale from "Strongly agree" to "Strongly disagree". There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Treatment Choice and Treatment Received | 1 week Post-Decision Aid, 1 month post-decision, & 3 months post-decision
  Treatment Choice will be assessed by asking participants to identify which treatment they chose. Using electronic health records, we will record the child's actual treatment in case of parental change of mind or misreport. A "better" score would be matching the treatment choice declaration with whichever treatment the electronic health record indicates that the patient received.
Control Preference Scale | 1 week post baseline, 1 week post decision aid, 1 month post-decision
  This scale assesses participants' desire to participate in Shared Decision Making. This scale is an adaptation of the Degner & Sloan's Control Preference Scale. It is a one item question that asks people if they want to make the decision alone, with their clinician, or have their clinician make it. There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Acceptability of the Decision Aid | 1 week post decision aid
  This will be assessed with 5 questions. Participants will be asked questions about if they used the decision aid (DA) before their appointment or during their appointment, their likelihood to recommend the DA, the amount of information presented, and if the DA seemed biased. There is no "better" or more correct answer; it is up to the patient's opinion.
Consultation Quality | 1 week post baseline, 3 months post decision.
  2 items measuring the quality of consultation. One is asking the participant to rate their usefulness of consultation on a 7 point Likert scale that ranges from 0=not at all useful to 6=very useful. The second is asking the participant if the clinician encouraged any certain treatment. There is no "better" answer, as these are opinions.
SF-12 | 1 week post Baseline, 3 months post decision
  The 12-Item Short Form Health Survey (SF-12) is a validated scale measuring the participant's health that was designed to reduce respondent burden while achieving minimum standards of precision for purposes of group comparisons involving multiple health dimensions. Answers are given on a 5 point Likert scale ranging from 1=excellent to 5=poor for three of the questions (lower scores are better); answers are given in a dichotomous (yes/no) format for four of the questions ("yes" is better); answers are given on a 6 point Likert scale ranging from 1=all of the time to 6=none of the time for three of the questions (lower scores are better); answers are given in a trichotomous format (yes, limited a little; yes, limited a lot; no, not limited at all) for the remaining two questions ("no" is the better answer).
Use of Information Sources | 1 week post decision aid
  Participants indicate whether they consulted any of 10 sources of health information. Of these 10 sources, 2 ask about personal relationships (i.e., relatives and friends), 3 had their roots in massmedia (i.e., exposure to television/movies, magazines, and books about CHD), and 2 were educational/research-based (i.e., scientific journals/research papers and the internet). The remaining 3 sources included providers, support groups, and other parents who have a child with CHD. Answers are in a 5 point Likert scale ranging from 1=never to 5=a great deal. There is no right or wrong answer; it is up to patient preference, so no answer indicates a "better" than another.
Impact of a Child with Congenital Anomalies on Parents | 1 month post decision, 3 months post decision
  ICCAP is a validated questionnaire developed to assess the impact of giving birth to a child with severe anatomical congenital anomalies on parental quality of life as a result of early stress. There are 32 questions: 4 ask about contact with caregivers, 6 ask about support from social network, 5 ask about partner relationships, 4 ask about the participant's state of mind, and the remaining 13 ask about fear and anxiety. Answers range on a 4 point Likert scale that ranges from 1=strongly disagree to 4=strongly agree, with a "not applicable". With the first three categories (contact with caregivers, social network, and partner relationships), a higher score is a "better" score; the remaining two categories (state of mind and fear/anxiety) are reverse-scored, so a lower score is "better".

CONTACTS AND LOCATIONS:
Overall Officials: Angela Fagerlin, PhD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Primary Children's Hospital Fetal and Pediatric Cardiology Clinics or Cardiac or Neonatal Intensive Care Units, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito M, Nakajima S, Fujisawa D, Miyashita M, Kim Y, Shear MK, Ghesquiere A, Wall MM. Brief measure for screening complicated grief: reliability and discriminant validity. PLoS One. 2012;7(2):e31209. doi: 10.1371/journal.pone.0031209. Epub 2012 Feb 14. PMID 22348057
- [Background] Prigerson HG, Maciejewski PK, Reynolds CF 3rd, Bierhals AJ, Newsom JT, Fasiczka A, Frank E, Doman J, Miller M. Inventory of Complicated Grief: a scale to measure maladaptive symptoms of loss. Psychiatry Res. 1995 Nov 29;59(1-2):65-79. doi: 10.1016/0165-1781(95)02757-2. PMID 8771222
- [Background] Toedter LJ, Lasker JN, Alhadeff JM. The Perinatal Grief Scale: development and initial validation. Am J Orthopsychiatry. 1988 Jul;58(3):435-49. doi: 10.1111/j.1939-0025.1988.tb01604.x. PMID 3407734
- [Background] Allen KA. Parental decision-making for medically complex infants and children: an integrated literature review. Int J Nurs Stud. 2014 Sep;51(9):1289-304. doi: 10.1016/j.ijnurstu.2014.02.003. Epub 2014 Feb 20. PMID 24636443
- [Background] Coulter A, Stilwell D, Kryworuchko J, Mullen PD, Ng CJ, van der Weijden T. A systematic development process for patient decision aids. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S2. doi: 10.1186/1472-6947-13-S2-S2. Epub 2013 Nov 29. PMID 24625093
- [Background] Fagerlin A, Pignone M, Abhyankar P, Col N, Feldman-Stewart D, Gavaruzzi T, Kryworuchko J, Levin CA, Pieterse AH, Reyna V, Stiggelbout A, Scherer LD, Wills C, Witteman HO. Clarifying values: an updated review. BMC Med Inform Decis Mak. 2013;13 Suppl 2(Suppl 2):S8. doi: 10.1186/1472-6947-13-S2-S8. Epub 2013 Nov 29. PMID 24625261
- [Background] Adams RC, Levy SE; COUNCIL ON CHILDREN WITH DISABILITIES. Shared Decision-Making and Children With Disabilities: Pathways to Consensus. Pediatrics. 2017 Jun;139(6):e20170956. doi: 10.1542/peds.2017-0956. PMID 28562298
- [Background] Neubauer K, Williams EP, Donohue PK, Boss RD. Communication and decision-making regarding children with critical cardiac disease: a systematic review of family preferences. Cardiol Young. 2018 Oct;28(10):1088-1092. doi: 10.1017/S1047951118001233. Epub 2018 Jul 31. PMID 30062980
- [Background] Kavanaugh K, Moro TT, Savage T, Mehendale R. Enacting a theory of caring to recruit and retain vulnerable participants for sensitive research. Res Nurs Health. 2006 Jun;29(3):244-52. doi: 10.1002/nur.20134. PMID 16676343
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] O'Connor AM. Validation of a decisional conflict scale. Med Decis Making. 1995 Jan-Mar;15(1):25-30. doi: 10.1177/0272989X9501500105. PMID 7898294
- [Background] Zikmund-Fisher BJ, Smith DM, Ubel PA, Fagerlin A. Validation of the Subjective Numeracy Scale: effects of low numeracy on comprehension of risk communications and utility elicitations. Med Decis Making. 2007 Sep-Oct;27(5):663-71. doi: 10.1177/0272989X07303824. Epub 2007 Jul 24. PMID 17652180
- [Background] Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. Patient Educ Couns. 2010 Jan;78(1):130-3. doi: 10.1016/j.pec.2009.05.012. Epub 2009 Jun 26. PMID 19560303
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] Fagerlin A, Zikmund-Fisher BJ, Ubel PA, Jankovic A, Derry HA, Smith DM. Measuring numeracy without a math test: development of the Subjective Numeracy Scale. Med Decis Making. 2007 Sep-Oct;27(5):672-80. doi: 10.1177/0272989X07304449. Epub 2007 Jul 19. PMID 17641137
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Edwards A, Elwyn G, Hood K, Robling M, Atwell C, Holmes-Rovner M, Kinnersley P, Houston H, Russell I. The development of COMRADE--a patient-based outcome measure to evaluate the effectiveness of risk communication and treatment decision making in consultations. Patient Educ Couns. 2003 Jul;50(3):311-22. doi: 10.1016/s0738-3991(03)00055-7. PMID 12900105
- [Background] Bekker HL, Hewison J, Thornton JG. Applying decision analysis to facilitate informed decision making about prenatal diagnosis for Down syndrome: a randomised controlled trial. Prenat Diagn. 2004 Apr;24(4):265-75. doi: 10.1002/pd.851. PMID 15065100
- [Background] Mazer P, Gischler SJ, Koot HM, Tibboel D, van Dijk M, Duivenvoorden HJ. Impact of a child with congenital anomalies on parents (ICCAP) questionnaire; a psychometric analysis. Health Qual Life Outcomes. 2008 Nov 23;6:102. doi: 10.1186/1477-7525-6-102. PMID 19025612
- [Derived] Delaney RK, Pinto NM, Ozanne EM, Stark LA, Pershing ML, Thorpe A, Witteman HO, Thokala P, Lambert LM, Hansen LM, Greene TH, Fagerlin A. Study protocol for a randomised clinical trial of a decision aid and values clarification method for parents of a fetus or neonate diagnosed with a life-threatening congenital heart defect. BMJ Open. 2021 Dec 10;11(12):e055455. doi: 10.1136/bmjopen-2021-055455. PMID 34893487